CLINICAL TRIAL: NCT01150266
Title: Alteplase for Waking Onset STROKE
Brief Title: Study for the Use of Alteplase in Patients Who Awaken With Stroke
Acronym: AWOKE
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Scripps Health (Other)
Responsible Party: Principal Investigator, Thomas M Hemmen, Director, UCSD Stroke Center, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AWOKE; 5P50NS044148 (NIH)
Record Dates: First submitted 2010-06-23; First posted 2010-06-24 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Ischemic Stroke
Keywords: stroke; ischemia; thrombolysis; thrombolytics; tPA; rt-PA; t-PA; Activase®; Alteplase; wake-up stroke; waking onset stroke; sleep
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alteplase (Experimental): Alteplase 0.9mg/kg (maximum 90mg), 10% IV bolus over 1 minute and the remainder over one hour infusion in patients with ischemic stroke after awaking.
  Interventions: Drug: Alteplase (tPA)

INTERVENTIONS:
Drug: Alteplase (tPA) — 0.9mg/KG (maximum 90mg), 10% bolus over one minutes, remainder over one hour.
  Other Names: Activase®; rt-PA; t-PA; tPA

SUMMARY:
This is a pilot study of thrombolytic therapy in patients with ischemic stroke who present with stroke symptoms upon awakening.

DETAILED DESCRIPTION:
Patients with ischemic stroke are currently only eligible for the treatment with intravenous thrombolysis if the stroke is diagnosed within 4.5 hours from known onset of symptoms.

Many patients awaken with stroke and are excluded from this therapy, following current guidelines.

Patients who suffer from a stroke just before or after waking up may be candidates for thrombolysis and our study will use advanced neuroimaging to select those patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥22
2. Stroke upon awakening
3. Measurable deficit by NIHSS
4. No deficit before sleep or last seen normal before to sleep
5. Head CT with no evidence of intracranial hemorrhage.
6. Able to receive IV t-PA treatment within 2.5 hrs after patient awoke with deficit.
7. Written informed consent signed and dated by the patient (or patient's authorized representative)
8. Core lesion: ASPECTS ≥7 on MRI-DWI, CTP-CBV or CTA source imaging.
9. Mismatch of at least 20% measured by CT CVB/MMT or DWI/TTP

Exclusion Criteria:

1. Stroke or serious head trauma within the preceding 3 months
2. Major surgery or serious trauma within 14 days
3. History of intracranial hemorrhage
4. Systolic blood pressure above 185 mm Hg or diastolic blood pressure above 110 mm Hg that is not controlled after aggressive measures.
5. Rapidly improving or minor symptoms
6. Symptoms suggestive of subarachnoid hemorrhage.
7. Gastrointestinal hemorrhage or urinary tract hemorrhage within the previous 21 days.
8. Arterial puncture at a non-compressible site within the previous 7 days
9. Seizure at the onset of stroke and considered the cause for the neurological symptom.
10. Patients who are taking anticoagulants or who had received heparin within the 48 hours preceding the onset of stroke and have an elevated partial-thromboplastin time, INR>1.7 or platelet counts below 100,000/mm3
11. Finger sticks glucose below 50 mg/dl (2.7 mmol/ Lt) or above 400 mg per deciliter (22.2 mmol/Lt) and considered the cause for the neurological symptom.
12. Active internal bleeding
13. Pregnancy in women of child-bearing potential (must have pregnancy test, urine or blood, prior to therapy).
14. Lumbar puncture within 7 days.
15. Known co-morbid conditions likely to complicate therapy or interfere with patient assessment, such us: heart failure stage 4, severe dementia, end-stage AIDS, pericarditis, cirrhosis or known cancer.
16. Unable to obtain CTA or perfusion brain studies (PWI or CTP)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Symptomatic Intracranial Hemorrhage | 0-72 hours
  sICH is defined as any confluent dense hematoma occupying greater than 30% of the infarcted area with substantial space occupying effect, or any brain hemorrhage outside the infarcted area that occurs within 72 hours of tPA treatment and is associated with an increase of at least 4 points in the NIHSS.

SECONDARY OUTCOMES:
Modified Rankin Scale | 90 days
  A good outcome is defined as a modified Rankin Scale (mRS) of ≤1 or return to baseline mRS.
National Institutes of Health Stroke Scale (NIHSS) | 24 hours
  An improvement of the NIHSS is defined as a 4-point improvement in the NIHSS, or NIHSS 0 measured 24 hours after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

REFERENCES:
- See also: UCSD Stroke Center — http://heartcenter.ucsd.edu/stroke